CLINICAL TRIAL: NCT07161258
Title: An Open-label, Single-arm Study to Evaluate Pharmacokinetics, Pharmacodynamic Effects, Safety and Tolerability of Fenebrutinib in Children and Adolescents With Relapsing Multiple Sclerosis
Brief Title: A Pharmacokinetics (PK), Pharmacodynamics (PD), Safety and Tolerability Study of Fenebrutinib in Children and Adolescents With Relapsing Multiple Sclerosis (RMS)
Acronym: FENerations1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN45847; 2024-519800-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Pediatric multiple sclerosis; Pediatric MS; Children MS; Children multiple sclerosis; Adolescent multiple sclerosis; Pediatric fenebrutinib
MeSH Terms: interventions — fenebrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fenebrutinib (Experimental): Participants will receive fenebrutinib orally.
  Interventions: Drug: Fenebrutinib

INTERVENTIONS:
Drug: Fenebrutinib — Fenebrutinib will be administered orally.

SUMMARY:
This open label, single arm study will evaluate the PK and PD effects of fenebrutinib in children and adolescents with RMS aged between 10 and < 18 years.

This study consists of a Dose Exploration Period and an Optional Extension Period. Eligible participants may choose to continue treatment with fenebrutinib in the optional extension period after completing the dose exploration period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RMS in accordance with the International Pediatric Multiple Sclerosis Study Group (IPMSSG) criteria for pediatric MS, Version 2012, and the revised 2017 McDonald Criteria and one or more of the following: at least one MS relapse during the previous year or two MS relapses in the previous 2 years or evidence of at least one Gd enhancing lesion on MRI within 6 month
* Expanded Disability Status Scale (EDSS) at screening from 0 to 5.5 points, inclusive
* Children and adolescents must have received all childhood vaccinations as per local/national recommendations for childhood vaccination against infectious diseases

Exclusion Criteria:

* A diagnosis of primary progressive multiple sclerosis (PPMS) or non-active secondary progressive multiple sclerosis (SPMS)
* Co-morbid Conditions:
* Potentially confounding neurological, somatic, or metabolic disorders
* Current clinically significant psychiatric or medical illness
* History of cancer, transplants, or bleeding disorders
* Inability to complete an MRI scan or get gadolinium
* Abnormal liver function tests or blood counts
* Peripheral venous access that precludes venous blood sampling as required per study protocol
* Sensitivity or intolerance to any ingredient (including excipients) of fenebrutinib tablets
* Active, recurrent, or chronic infections
* Recent or anticipated use of prohibited medications/treatments:
* Certain disease-modifying therapy (DMT) and other immunosuppressants
* Drugs interacting with fenebrutinib (Cytochrome P450 3A4 [CYP3A4] inhibitors)
* Any other investigational therapy, anticoagulants, certain vaccines

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2029-02-13 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Fenebrutinib | Up to Week 96
Total Number of New T1 Gadolinium (Gd)-Enhancing Lesions on Brain Observed Through Magnetic Resonance Imaging (MRI) Scans | At Week 12

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately 100 weeks
Percentage of Participants With Suicidal Ideation (SI) or Behavior, as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately 100 weeks
  The C-SSRS is an interview-based instrument used to assess baseline incidence of SI and behavior. The assessment includes yes/no (0/1) responses for 5 questions, each related to SI.
Change From Baseline in Vital Signs - Pulse Rate | Baseline up to approximately 100 Weeks
Change From Baseline in Vital Signs - Blood Pressure | Baseline up to approximately 100 Weeks
Change From Baseline in Single 12-lead Electrocardiogram (ECG) Parameter - QTc Interval | Baseline up to approximately 100 Weeks
Change From Baseline in Single 12-lead ECG Parameter - PR Interval | Baseline up to approximately 100 Weeks
Change from Baseline in Clinical Laboratory Test Results - Alanine Aminotransferase (ALT) | Baseline up to approximately 100 Weeks
Change from Baseline in Clinical Laboratory Test Results - Aspartate Aminotransferase (AST) | Baseline up to approximately 100 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Argentina (2):
  - INECO Neurociencias Orono, Rosario, Santa Fe Province
  - Sanatorio del Sur S.A., San Miguel de Tucumán
- Brazil (4):
  - L2IP ?Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - Instituto de Neurologia de Curitiba - Hospital Ecoville, Curitiba, Paraná
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul NPCR, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Clinicas - CPCLIN, São Paulo, São Paulo
- Mexico (2):
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
- Portugal (2):
  - Centro Clnico Acadmico - Braga, Associao (2CA-Braga), Braga
  - Unidade Local de Saude de Coimbra E P E, Coimbra
- Spain (3):
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- CNE of Lviv Reg Clin Hospital Dept of Neurology D.Halytskyi Lviv NMU, Lviv, KIEV Governorate, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing